CLINICAL TRIAL: NCT06934304
Title: Randomized Controlled Study on Patient Preoperative Preparedness and Satisfaction Using a Redesigned Handout for Robotic Sacrocolpopexy
Brief Title: The Impact of a Redesigned Handout for Robotic Sacrocolpopexy on Patient Preoperative Preparedness and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of Texas, Southwestern Medical Center at Dallas (Other)
Responsible Party: Principal Investigator, Christine Herforth, Urology Fellow, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STU-2022-0305
Record Dates: First submitted 2025-04-04; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Pelvic Organ Prolapse; Patient Satisfaction
Keywords: Robotic sacrocolpopexy handout study
MeSH Terms: conditions — Pelvic Organ Prolapse; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Old preoperative handout (Placebo Comparator): Standard or old preoperative handout for robotic sacrocolpopexy was based off of the handout for robotic sacrocolpopexy from the American Urogynecologic Society
  Interventions: Other: old preoperative handout
- New preoperative handout (Experimental): A new preoperative handout for robotic sacrocolpopexy was designed by changing the old preoperative handout such that it was written at a lower grade reading level and provided more perioperative details
  Interventions: Other: new preoperative handout

INTERVENTIONS:
Other: new preoperative handout — A new preoperative handout for robotic sacrocolpopexy was designed at a lower reading level and providing more perioperative details
  Arms: New preoperative handout
Other: old preoperative handout — The old or standard preoperative handout for robotic sacrocolpopexy
  Arms: Old preoperative handout

SUMMARY:
The goal of this clinical trial is to learn if a new preoperative handout for patients undergoing robotic sacrocolpopexy will improve patient sense of preparedness and satisfaction in comparison to the previously used handout. The main questions it aims to answer are:

* Does the new preoperative handout for patients undergoing robotic sacrocolpopexy improve patient preparedness and satisfaction?
* Will the new preoperative handout for patients undergoing robotic sacrocolpopexy impact postoperative queries in the form of phone calls and messages to the clinic?

Participants will:

* Receive routine counseling regarding robotic sacrocolpopexy from their surgeon
* Be randomized to the new or old preoperative handout
* Undergo robotic sacrocolpopexy
* Complete a questionnaire at their 4 week postoperative follow up visit regarding their sense of preparedness for surgery and overall satisfaction

ELIGIBILITY:
Inclusion Criteria:

* women who were to undergo robotic sacrocolpopexy with or without supracervical hysterectomy, rectopexy, salpingectomy, urinary incontinence procedures, or other minor procedures.

Exclusion Criteria:

* patients unable to provide informed consent, those undergoing other concomitant major abdominal surgeries, patients less than 18 years old, pregnant patients, non-English speaking patients, and patients planning postoperative follow up at an outside facility.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Patient preparedness | Assessed at the postoperative visit 4 to 6 weeks after srugery
  Patients sense of preparedness for robotic sacrocolpopexy was measured with a series of 5 point Likert style questions (ranging strongly disagree to strongly agree). Specifically, patients were asked how satisfied the were with 1) information provided by their surgeon, 2) time spent with the patient preparing them for surgery, 3) overall sense of sense of preparedness.

SECONDARY OUTCOMES:
patient satisfaction | 4 week postoperatively
  patient satisfaction for their overall experience undergoing robotic was assessed using a 5 point patient score. Scores ranged from extremely dissatisfied to extremely satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No